CLINICAL TRIAL: NCT05886400
Title: The Effects of Environmental Distractions on SCAT6 Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Keisuke Kawata, Associate Professor, Indiana University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: 18810
Record Dates: First submitted 2023-05-23; First posted 2023-06-02 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Concussion, Brain; Mild Traumatic Brain Injury
Keywords: Standardized Concussion Assessment Tool; Modified Balance Error Scoring System; Sports Participation
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Distracted (Experimental): Visual and audio distraction via sports video clips or a game will be playing during the testing session.
  Interventions: Other: SCAT6; Other: Visual/ Auditory Distraction
- Not Distracted (Sham Comparator): No visual or auditory distractions will be used during testing session. Testing area will be in a controlled environment.
  Interventions: Other: SCAT6

INTERVENTIONS:
Other: SCAT6 — The SCAT6 is a standardized assessment tool to diagnose a concussion. This tool will be used for the experiment utilizing the 6th edition to recreate the methods used in an athletic situation. The SCAT6 is broken down into multiple subtests to focus on specific aspects of a person's wellbeing that could be affected by a possible concussion. The assessments are created to measure an athlete's subjectively experienced symptoms, cognitive functioning and balance and postural stability (mBESS).
  Other Names: Standardized Concussion Assessment Tool
Other: Visual/ Auditory Distraction — The purpose of this study is to examine the effect of environmental distractions on one's ability to complete the SCAT6. The environmental distractions will be visual and auditory by playing a sports event or sports clips during the completion of the assessment. The goal of this is to simulate the distraction of a sideline like a SCAT6 is typically used within athletic training.
  Arms: Distracted

SUMMARY:
The purpose of this study is to assess the effects of visual and auditory distractions on SCAT5 scores. The study is designed to identify the effects of about 80 participants completing the SCAT5 in college-aged athletes. All participants will perform the same tasks in two settings (distracted and non-distracted). The central hypothesis is that there will be a significant association between distractions and a lower score on the SCAT5. The cognitive screening, neurological screen, and mBESS should showcase a decrease scores during the distracted environment.

DETAILED DESCRIPTION:
The researchers will use a randomized controlled trial design and recruit participants on a first-come, first-serve basis for the study. This crossover design will consist of two groups. The two groups are; distracted and non-distracted. The study will consist of two time points in an 8-day period.

After the initial recruitment email and enrollment questionnaire, those who are eligible for the study will be randomly assigned to begin in one of the two groups. The researchers will include a self-reported health questionnaire to obtain demographic information. The information includes age, sex, race/ ethnicity, years of athletic experience, number of previous concussions, favorite sports (with gender and level) to watch, and an assessment of other neurological conditions to screen participants' eligibility. Participants who meet the inclusion criteria and are free of exclusionary factors will advance to the consent forms and testing procedures. Consent forms will be filled out via Qualtrics.

Symptom Evaluation:

The symptom evaluation assesses severity and presence of symptoms. The symptom evaluation requires participants to self-report a total of 22 on a 7-point Likert scale ranging from 0 (none) to 7 (severe). Participants will be instructed to truthfully report their symptoms by circling their scores. Symptom scores will be manually transferred to an Excel spreadsheet for future analyses.

Cognitive Screening:

The cognitive screening portion of the SCAT5 is adapted from the standardized assessment of concussion (SAC). This section consists of orientation questions (like what day is it?) followed by immediate memory. Immediate memory consists of 5-item list of words presented to the participant three times and the participants are asked to recite the words back in any order. After the immediate memory assessment concentration is assessed using the digits backwards and months in reverse order tests. The digits backwards test starts with the participants being given a series of 3 numbers and asked to repeat them in reverse order, the test progresses up to 6 numbers. The test is discontinued after 2 consecutive incorrect answers. The months backwards test requires participants to recite the months of the year in reverse order. Following the months backwards the participant is asked to give as many words from the 5-item list as they can remember.

Neurological Screen :

The neurological screen is a brief series of questions assessing neurological function of the participant. This screen consists of participants ability to read out loud and follow instructions, perform full pain-free passive range of motion, vertical and horizontal eye movement (without moving the head), and complete tandem gait. Tandem gait requires participant to stand with their feet together (footwear off), they are instructed to walk as quickly and accurately as possible along the line in front of them maintaining an alternating foot heel to toe gait. The test is discontinued if the participant steps off of the line or does not maintain contact between heel and toe of opposite feet.

Modified Balance Error Scoring System (mBESS):

The balance testing is a modified version of the Balance Error Scoring System. The test consists of 20 second trials for 3 separate stances. The stances consist of double leg balance, single leg balance (non-dominant leg) and a tandem stance. Each stance will be performed with the participants hands on their hips and eyes closed. The scoring for this assessment is counted for every error that occurs during each stance. The errors include hands off hips, opening eyes, step/stumble/fall, moving hips into greater than 30 degrees of abduction, lifting heel or forefoot and staying out of position for greater than 5 seconds. Maximum number of errors is 10. If the participant cannot maintain position for a minimum of 5 seconds the test is discontinued and an automatic error score of 10 is given.

ELIGIBILITY:
Inclusion Criteria:

* Previous athletic experience beginning at or after the age of 12

Exclusion Criteria:

* Diagnosed with a neurological condition (including epilepsy, stroke, seizures)
* Have had a concussion within the past 6 months (diagnosed or undiagnosed)
* have not participated in sport

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Significant association between visual and auditory distractions and the outcomes of the Standardized Concussion Assessment Tool (SCAT6) assessment | Completion of both environments to analyze the differences in scores will be completed on day 8.
  Scores on the SCAT6 will differ between the control and non-distracted environment. Specifically for the main portion of the SCAT6 the orientation, immediate memory, concentration, and delayed recall scores will be compiled. Scores can be a minimum of 0 and a maximum of 50. A higher score indicates better performance while a lower score indicates worse performance.

SECONDARY OUTCOMES:
Symptom list | Completion of both environments to analyze the differences in scores will be completed on day 8.
  Scores on the symptom list will not show differences between the control / non-distracted environment and experimental / distracted environment. The symptom list portion can have a minimum score of 0 for both the number of symptoms and severity of symptoms. It can have a maximum score of 22 for total number of symptoms and a maximum score of 132 for symptom severity. A lower score indicates a better outcome while a higher score indicates a worse outcome.
Modified Balance Error Scoring System (mBESS) | Completion of both environments to analyze the differences in scores will be completed on day 8.
  Scores on the SCAT6 will differ between the control and non-distracted environment. During the mBESS the minimum score is a 0 and the maximum score is 30. A lower score indicates better performance while a higher score indicates worse performance.

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University School of Public Health, Bloomington, Indiana, United States

IPD SHARING:
Plan to Share IPD: No
All study data will be included in publications.

REFERENCES:
- [Background] Taylor CA, Bell JM, Breiding MJ, Xu L. Traumatic Brain Injury-Related Emergency Department Visits, Hospitalizations, and Deaths - United States, 2007 and 2013. MMWR Surveill Summ. 2017 Mar 17;66(9):1-16. doi: 10.15585/mmwr.ss6609a1. PMID 28301451
- [Background] Laker SR. Epidemiology of concussion and mild traumatic brain injury. PM R. 2011 Oct;3(10 Suppl 2):S354-8. doi: 10.1016/j.pmrj.2011.07.017. PMID 22035677
- [Background] McCrory P, Meeuwisse W, Johnston K, Dvorak J, Aubry M, Molloy M, Cantu R. Consensus statement on concussion in sport: the 3rd International Conference on Concussion in Sport held in Zurich, November 2008. J Athl Train. 2009 Jul-Aug;44(4):434-48. doi: 10.4085/1062-6050-44.4.434. No abstract available. PMID 19593427
- [Background] Teel EF, Register-Mihalik JK, Appelbaum LG, Battaglini CL, Carneiro KA, Guskiewicz KM, Marshall SW, Mihalik JP. Randomized Controlled Trial Evaluating Aerobic Training and Common Sport-Related Concussion Outcomes in Healthy Participants. J Athl Train. 2018 Dec;53(12):1156-1165. doi: 10.4085/1062-6050-7-18. Epub 2018 Dec 18. PMID 30562056
- [Background] Hanninen T, Parkkari J, Howell DR, Palola V, Seppanen A, Tuominen M, Iverson GL, Luoto TM. Reliability of the Sport Concussion Assessment Tool 5 baseline testing: A 2-week test-retest study. J Sci Med Sport. 2021 Feb;24(2):129-134. doi: 10.1016/j.jsams.2020.07.014. Epub 2020 Aug 5. PMID 32868203
- [Background] Echemendia RJ, Meeuwisse W, McCrory P, Davis GA, Putukian M, Leddy J, Makdissi M, Sullivan SJ, Broglio SP, Raftery M, Schneider K, Kissick J, McCrea M, Dvorak J, Sills AK, Aubry M, Engebretsen L, Loosemore M, Fuller G, Kutcher J, Ellenbogen R, Guskiewicz K, Patricios J, Herring S. The Sport Concussion Assessment Tool 5th Edition (SCAT5): Background and rationale. Br J Sports Med. 2017 Jun;51(11):848-850. doi: 10.1136/bjsports-2017-097506. Epub 2017 Apr 26. PMID 28446453
- [Background] Yengo-Kahn AM, Hale AT, Zalneraitis BH, Zuckerman SL, Sills AK, Solomon GS. The Sport Concussion Assessment Tool: a systematic review. Neurosurg Focus. 2016 Apr;40(4):E6. doi: 10.3171/2016.1.FOCUS15611. PMID 27032923
- [Background] Black AM, Miutz LN, Kv VW, Schneider KJ, Yeates KO, Emery CA. Baseline Performance of High School Rugby Players on the Sport Concussion Assessment Tool 5. J Athl Train. 2020 Feb;55(2):116-123. doi: 10.4085/1062-6050-123-19. Epub 2020 Jan 9. PMID 31917599
- [Background] Iverson GL, Howell DR, Van Patten R, Bloomfield P, Gardner AJ. Sport Concussion Assessment Tool-5th Edition (SCAT5): Normative Reference Values for the National Rugby League Women's Premiership. Front Sports Act Living. 2021 May 26;3:653743. doi: 10.3389/fspor.2021.653743. eCollection 2021. PMID 34124655
- [Background] Petit KM, Savage JL, Bretzin AC, Anderson M, Covassin T. The Sport Concussion Assessment Tool-5 (SCAT5): Baseline Assessments in NCAA Division I Collegiate Student-Athletes. Int J Exerc Sci. 2020 Aug 1;13(3):1143-1155. doi: 10.70252/SUJD2658. eCollection 2020. PMID 32922635
- [Background] Bland DC, Zampieri C, Damiano DL. Effectiveness of physical therapy for improving gait and balance in individuals with traumatic brain injury: a systematic review. Brain Inj. 2011;25(7-8):664-79. doi: 10.3109/02699052.2011.576306. Epub 2011 May 11. PMID 21561297
- [Background] Dessy AM, Yuk FJ, Maniya AY, Gometz A, Rasouli JJ, Lovell MR, Choudhri TF. Review of Assessment Scales for Diagnosing and Monitoring Sports-related Concussion. Cureus. 2017 Dec 7;9(12):e1922. doi: 10.7759/cureus.1922. PMID 29456902
- [Background] West TA, Marion DW. Current recommendations for the diagnosis and treatment of concussion in sport: a comparison of three new guidelines. J Neurotrauma. 2014 Jan 15;31(2):159-68. doi: 10.1089/neu.2013.3031. Epub 2013 Oct 16. PMID 23879529
- [Background] Mistry DA, Rainer TH. Concussion assessment in the emergency department: a preliminary study for a quality improvement project. BMJ Open Sport Exerc Med. 2018 Dec 27;4(1):e000445. doi: 10.1136/bmjsem-2018-000445. eCollection 2018. PMID 30687512
- [Background] Lempke LB, Schmidt JD, Lynall RC. Athletic Trainers' Concussion-Assessment and Concussion-Management Practices: An Update. J Athl Train. 2020 Jan;55(1):17-26. doi: 10.4085/1062-6050-322-18. Epub 2019 Dec 19. PMID 31855075
- [Background] Shanley E, Thigpen CA, Chapman CG, Thorpe J, Gilliland RG, Sease WF. Athletic Trainers' Effect on Population Health: Improving Access to and Quality of Care. J Athl Train. 2019 Feb;54(2):124-132. doi: 10.4085/1062-6050-219-17. Epub 2018 Nov 21. PMID 30461294
- [Background] Starling AJ, Leong DF, Bogle JM, Vargas BB. Variability of the modified Balance Error Scoring System at baseline using objective and subjective balance measures. Concussion. 2015 Aug 6;1(1):CNC5. doi: 10.2217/cnc.15.5. eCollection 2016 Mar. PMID 30202550
- [Background] Guskiewicz KM. Balance assessment in the management of sport-related concussion. Clin Sports Med. 2011 Jan;30(1):89-102, ix. doi: 10.1016/j.csm.2010.09.004. PMID 21074084
- [Background] Ruhe A, Fejer R, Gansslen A, Klein W. Assessing postural stability in the concussed athlete: what to do, what to expect, and when. Sports Health. 2014 Sep;6(5):427-33. doi: 10.1177/1941738114541238. PMID 25177420
- [Background] Bell DR, Guskiewicz KM, Clark MA, Padua DA. Systematic review of the balance error scoring system. Sports Health. 2011 May;3(3):287-95. doi: 10.1177/1941738111403122. PMID 23016020
- [Background] Quatman-Yates C, Hugentobler J, Ammon R, Mwase N, Kurowski B, Myer GD. The utility of the balance error scoring system for mild brain injury assessments in children and adolescents. Phys Sportsmed. 2014 Sep;42(3):32-8. doi: 10.3810/psm.2014.09.2073. PMID 25295764
- [Background] Silverberg ND, Iaccarino MA, Panenka WJ, Iverson GL, McCulloch KL, Dams-O'Connor K, Reed N, McCrea M; American Congress of Rehabilitation Medicine Brain Injury Interdisciplinary Special Interest Group Mild TBI Task Force. Management of Concussion and Mild Traumatic Brain Injury: A Synthesis of Practice Guidelines. Arch Phys Med Rehabil. 2020 Feb;101(2):382-393. doi: 10.1016/j.apmr.2019.10.179. Epub 2019 Oct 23. PMID 31654620
- [Background] Broglio SP, Cantu RC, Gioia GA, Guskiewicz KM, Kutcher J, Palm M, Valovich McLeod TC; National Athletic Trainer's Association. National Athletic Trainers' Association position statement: management of sport concussion. J Athl Train. 2014 Mar-Apr;49(2):245-65. doi: 10.4085/1062-6050-49.1.07. Epub 2014 Mar 7. PMID 24601910
- [Background] King D, Brughelli M, Hume P, Gissane C. Assessment, management and knowledge of sport-related concussion: systematic review. Sports Med. 2014 Apr;44(4):449-71. doi: 10.1007/s40279-013-0134-x. PMID 24403125
- [Background] Scorza KA, Cole W. Current Concepts in Concussion: Initial Evaluation and Management. Am Fam Physician. 2019 Apr 1;99(7):426-434. PMID 30932451
- [Background] Harmon KG, Drezner JA, Gammons M, Guskiewicz KM, Halstead M, Herring SA, Kutcher JS, Pana A, Putukian M, Roberts WO. American Medical Society for Sports Medicine position statement: concussion in sport. Br J Sports Med. 2013 Jan;47(1):15-26. doi: 10.1136/bjsports-2012-091941. PMID 23243113
- [Background] Miller PC, Hall EE, Bailey EK. The Influence of Various Distraction Stimuli on Affective Responses during Recumbent Cycle Ergometry. Sports (Basel). 2016 Mar 23;4(2):21. doi: 10.3390/sports4020021. PMID 29910269
- [Background] Flanagan SR. Invited Commentary on "Centers for Disease Control and Prevention Report to Congress: Traumatic Brain Injury in the United States: Epidemiology and Rehabilitation". Arch Phys Med Rehabil. 2015 Oct;96(10):1753-5. doi: 10.1016/j.apmr.2015.07.001. Epub 2015 Jul 14. PMID 26184889